CLINICAL TRIAL: NCT05237752
Title: A Phase Ib/II, Double-blind, Placebo-controlled Study to Evaluate the Safety and Efficacy of a Single Dose of LG00034053 Administered by Intra-articular Injection in Patients With Knee Osteoarthritis
Brief Title: A Phase Ib/II Clinical Trial to Evaluate the Safety and Efficacy of LG00034053 in Patients With Knee OA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: LG Chem (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LG-CSCL004
Record Dates: First submitted 2021-11-17; First posted 2022-02-14 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LG00034053 (Experimental): White to slightly brown powder, dosage (6mg, 15mg, 45mg; dose escalation design), single dose administration
  Interventions: Drug: LG00034053
- Placebo (Placebo Comparator): Clear liquid, single dose administration
  Interventions: Drug: LG00034053

INTERVENTIONS:
Drug: LG00034053 — a pan-caspase inhibitor, as a therapeutic agent of osteoarthritis

SUMMARY:
This study is a multi-center, randomized, placebo-controlled, double-blind clinical study, consisting of Part 1 (Phase 1b) in a sequential, dose-escalating design and Part 2 (Phase 2) in a parallel design.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with primary osteoarthritis of the knee according to the ACR clinical criteria, with Kellgren-Lawrence grade 2 to 3 in the corresponding knee as determined in the X-ray test
* Patients with pain in the index knee requiring NSAIDs or analgesics which sustained for at least 6 months
* Patients with a score of ≥ 4 and ≤ 9 in response to question 1 (walking pain) on the WOMAC pain subscale (11-point NRS)
* Patients with the subtotal score of ≥ 20 and ≤ 45 on the WOMAC pain subscale (11- point NRS)
* Patients with BMI at or below 40 kg/m2

Exclusion Criteria:

* Patients with chronic pain requiring continuous treatment
* Patients with rheumatoid arthritis or other inflammatory arthritis
* Patients with skin disorders at the administration site
* Patients with clinically significant renal or cardiovascular disease or those with suspected SARS-CoV-2 infection
* Patients in a medical condition which may affect the efficacy and/or safety assessment
* Patients with Kellgren-Lawrence grade 4 in the contralateral knee
* Patients with tense effusion
* Patients having administered an opioid analgesic/ other analgesic/health functional foods, single dose of IA injection within a certain period prior to drug administration
* Patients having undergone knee replacement

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2022-04-27 (Actual); Primary Completion 2023-12-19 (Actual); Study Completion 2024-03-11 (Actual)

PRIMARY OUTCOMES:
Changes in WOMAC (Western Ontario and McMaster Universities Arthritis Index) (11-point NRS) pain score from baseline to time point | week 12
  Change of WOMAC (11-point NRS) pain score from baseline to Week 12
  - a total of 5 questions, each question's score is as below Mininum : 0 (no pain) Maximum : 10 (extreme pain) Higher score means worse outcome

SECONDARY OUTCOMES:
Change in WOMAC score from baseline to time point | week 1 ~ week 24
  Change of WOMAC (11-point NRS) score
  1. WOMAC pain score (except week 12)
  2. WOMAC function, stiffness, total score
     * function (17 questions, scores are 0 to 170)
     * stiffness (2 questions, scores are 0 to 20)
     * total score: pain + function + stiffness = 240 at maximum Higher score means worse outcome
Weekly mean of the average daily pain intensity score (11-point NRS) from baseline to time point | week 1 ~ week 24
  Change in weekly mean of average daily pain intensity score (11-point NRS)
  - 0 (no pain) to 10 (pain as bad as you can imagine)

CONTACTS AND LOCATIONS:
Locations (2):
- Emeritus Research, Camberwell, Australia
- The Catholic Univ. of Korea Seoul St. Mary's Hospital, Seoul, South Korea